CLINICAL TRIAL: NCT03698942
Title: A Retrospective, Observational, Case-Controlled, Multi-Reader, Multi-Case, Receiver Operating Characteristic (ROC) Study of Reader Performance When SoftVue Automated Breast Ultrasound (SV) and Digital Screening Mammography (DM) Are Combined, Compared to Screening Mammography Alone, in Asymptomatic Women With Heterogeneous or Extremely Dense Breast Parenchyma.
Brief Title: Delphinus SoftVue™ ROC Reader Study
Acronym: DMT SV RRS1
Status: Completed | Type: Observational
Sponsor: Delphinus Medical Technologies, Inc. (Industry)
Collaborators: University of Chicago (Other); Biostatistics Consulting, LLC (Unknown); Reed Technical Associates, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: DMT-2015.002
Record Dates: First submitted 2018-08-13; First posted 2018-10-09 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Breast Screening; Breast Imaging; SoftVue; Mammography; Ultrasound; Reader Study; ROC AUC; Breast Cancer Detection; Dense Breasts; Breast Density; Dense Breast Tissue; Dense Breast Parenchyma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Reading of Automated Breast Ultrasound in conjunction with Screening Mammography — Reader performance when SoftVue automated breast ultrasound (SV) and digital screening mammography (DM) are combined, compared to screening mammography alone.
  Other Names: Digital Screening Mammography with SoftVue Supplemental Screening Whole Breast Ultrasound

SUMMARY:
The purpose of this multi-reader, multi-case (MRMC) reader study is to evaluate reader performance when SoftVue™ automated breast ultrasound and screening mammography are combined, compared to screening mammography alone, in women with dense breast parenchyma. This includes obtaining information that can be used to properly plan, design, and power future ROC reader studies.

This reader study will include a minimum of 6 radiologist readers and an enriched sample of at least 100 breast screening or diagnostic cases to be selected from the library of images collected under Delphinus Protocol #DMT-2015.001 (NCT03257839). The reader study image case set will be enriched with cancer cases.

ELIGIBILITY:
Radiologists of any age, sex, race, ethnicity, or institutional affiliation may participate as study readers. All readers must meet the following Inclusion Criteria:

* Hold a current United States medical license
* Be American Board of Radiology Certified
* Be MQSA-qualified
* Be experienced in reading FFDM images on a monitor (softcopy)
* Be experienced in reading Breast Ultrasound images on a monitor (softcopy)
* Have completed a Financial Disclosure showing no Conflicts of Interest
* Have provided a current curriculum vitae (CV)
* Have provided a signed Readers' Agreement
* Have provided written Informed Consent

All qualified and confirmed readers will complete a multi-module SoftVue™ training program prior to their participation in a reading session for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Readers will evaluate mammography and SoftVue images acquired at study entry in protocol DMT 2015.001 and subsequently categorized into the following case types, in random order:
  * Cancer cases, confirmed by breast biopsy with at least one lesion determined to be malignant during participation
  * Non-Cancer cases including, but not limited to benign cases, confirmed by breast biopsy with no lesions determined to be malignant, or normal/negative screening or diagnostic imaging during participation
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
MRMC Analysis: ROC AUC | 8 Weeks
  Area under the ROC curve (AUC)

SECONDARY OUTCOMES:
Sensitivity and Specificity | 8 Weeks
  True Positive Rate and True Negative Rate

CONTACTS AND LOCATIONS:
Overall Officials: Yulei Jiang, Ph.D, Principal Investigator — University of Chicago; Mary Ellen Giger, Ph.D, Principal Investigator — Univeristy of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No